CLINICAL TRIAL: NCT00558246
Title: Multi-centre Study to Show Equivalence of Prineo (DERMABOND PROTAPE) to Intradermal Sutures for Skin Closure of Full-thickness Surgical Incisions Associated With Breast Procedures
Brief Title: Study of Prineo (Dermabond Protape) Versus Sutures in Breast Procedures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07CS003
Record Dates: First submitted 2007-11-09; First posted 2007-11-14 (Estimated); Results first posted 2012-07-19 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-06

CONDITIONS: Macromastia
Keywords: Breast Lift; Breast Reduction; Breast Reconstruction; Plastic Surgery; Skin Closure; Wound Healing; Dermabond
MeSH Terms: conditions — Gigantomastia | interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): On same patient, one breast is randomized to control and one breast is randomized to experimental arm. Patient is own control.
  Interventions: Device: Dermabond Protape (Prineo)
- II (Active Comparator): On same patient, one breast is randomized to control and one breast is randomized to experimental arm. Patient is own control.
  Interventions: Device: Suture

INTERVENTIONS:
Device: Dermabond Protape (Prineo) — cyanoacrylate and pressure sensitive adhesive mesh - topical skin adhesive
  Other Names: Prineo
  Arms: I
Device: Suture — Topical Suturing
  Other Names: Investigator selected the intradermal suture per standard local practice.
  Arms: II

SUMMARY:
This is a prospective, controlled, randomized, multi-center clinical study of up to 80 patients with full thickness surgical incisions associated with bi-lateral breast procedures. Breast procedures where symmetrical incisions of at least 15cm in length are planned for both breast (bilateral procedure) will be randomised to receive final skin closure of one breast with Prineo (DERMABOND PROTAPE) and the other with intradermal sutures (control). Patients will be evaluated post-operatively at 24 hours (± 6 hours), 7 days (± 1 day), 12 - 25 days, and 90 days (± 10 days).

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Be in good general health in the opinion of the Investigator with no conditions that would significantly impact wound healing as determined by medical history and review of recent concomitant medications;
* Require identical skin closure of full-thickness intersecting surgical incisions with a combined length of at least 15cm on each breast as part of elective breast procedures, requiring the placement of sutures in the superficial fascia and subcutaneous tissue to relieve skin tension prior to final skin closure;
* Be willing to follow instructions for incision care as instructed by the investigator, and refrain from swimming or soaking in a tub until suture removal occurs (during the first 12-25 days) of the study;
* Agree to return for all follow-up evaluations specified in this protocol [7 days (± 1 day), 12 - 25 days, and 90 days (± 10 days)], six (± 1 month) and twelve months (± 1 month)];
* Agree not to schedule any additional elective surgical procedures that involve an incision that is randomized for inclusion in this study, until their participation in this study is complete; and
* Sign the informed consent.

Exclusion Criteria:

* Have peripheral vascular disease;
* Have insulin dependent diabetes mellitus;
* Be known to have a blood clotting disorder;
* Be receiving antibiotic therapy for pre-existing condition or infection;
* Be known to be HIV-positive or otherwise immunocompromised;
* Have known personal or family history of keloid formation or hypertrophy;
* Be currently taking systemic steroids;
* Have known or suspected allergy or sensitivity to cyanoacrylate, formaldehyde, tapes or adhesives
* Have incision type or location known to have an incidence of cyanosis or other healing abnormalities; and
* Be participating in any current clinical trial of an investigational product or have participated in any clinical trial of an investigational product within 30 days of enrolment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Colquhoun, MD, Study Director — Pleiad Devices
Locations (5):
- UZ, Ghent, Belgium
- Germany (2):
  - Dreifaltigkeits-Krankenhaus, Cologne
  - Markus Krankenhaus, Frankfurt
- Akademikliniken, Stockholm, Sweden
- Mid Essex Hospital, Broomfield, Essex, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the genreal popluation of those undergoing elective, bilateral breast surgery.
Groups:
- Prineo and Suture: On same patient, one breast is randomized to control (intradermal sutures) and one breast is randomized to experimental arm (DERMABOND PROTAPE). Patient is own control. Protape is supplied as a single use mesh device with sufficient adhesive to saturate mesh. Sutures were not supplied.
Period: Overall Study
Arm/Group | Prineo and Suture
Started | 79
Completed | 79
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Prineo and Suture
Number analyzed (Participants) | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 78
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 10
  Germany | 47
  United Kingdom | 6
  Sweden | 16

OUTCOME MEASURES:

1. Primary Outcome: Continuous Apposition of the Skin Edges Without Wound Dehiscence or Re-closure as Measured by the Upper Limit of 95% Confidence Interval in Proportion of Successes for Each Groups.
Description: Equivalence was demonstrated if the upper limit of the 95% confidence interval (when subtracting the percentage of DERMABOND PROTAPE successful subjects from the percentage of INTRADERMAL SUTURE successful subjects) did not exceed 12 percent.
Time Frame: 12-25 days
Population: The primary analysis is based upon intent to treat population.
Measure: Number; unit: Participants
Groups:
- Prineo; Suture: On same patient, one breast is randomized to control and one breast is randomized to experimental arm. Patient is own control.
Arm/Group | Prineo | Suture
Number analyzed (Participants) | 79 | 79
Participants | 76 [-5.9 to 5.9] | 76 [-5.9 to 5.9]
Statistical Analysis 1: Comparison: Prineo vs Suture; Test type: Non-Inferiority or Equivalence — Equivalence is demonstrated if the upper limit of the 95% confidence interval (when subtracting the percentage of DERMABOND PROTAPE successful subjects from the percentage of INTRADERMAL SUTURE successful subjects) does not exceed 12%; p = 1.0000, McNemar; Differences in proportion of successes = 0, 95% CI 2-sided [-5.9 to 5.9] — The level of significance for statistical testing was 0.05 for this study

2. Secondary Outcome: Time (Minutes) Required to Close the Final Skin Layer
Description: Overall time required to close final skin layer on each breast.
Time Frame: Intraoperative
Population: The analysis is based upon the Intent to Treat population.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Prineo | Suture
Number analyzed (Participants) | 79 | 79
minutes | 2.56 (1.34) | 16.22 (6.41)
Statistical Analysis 1: Comparison: Prineo vs Suture; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

3. Secondary Outcome: Cosmetic Outcome
Description: Modified Hollander Cosmesis Scale overall outcome score in which a score of 0 corresponds to a good outcome versus a 1-6 to a poor outcome. The proportions of breasts with good outcomes were then compared to those with poor outcomes in each group.
  Reference: Hollander JE, Singer AJ, Valentine S, Thode HC Jr, Henry MC. Wound registry:development and validation. Ann Emerg Med. 1995;25:675-85.
Time Frame: 90 days post-procedure
Population: There were 60 participants who consented to and ultimately attended all follow-up visits for evaluation of cosmetic outcome.
Measure: Number; unit: Incisions with good outcome
Arm/Group | Prineo | Suture
Number analyzed (Participants) | 60 | 60
Incisions with good outcome | 49 | 49
Statistical Analysis 1: Comparison: Prineo vs Suture; Test type: Superiority or Other; p = 1.0000, McNemar

4. Secondary Outcome: Cosmetic Outcome
Description: as for outcome 3
Time Frame: 6 months
Population: There were 60 participants who completed all follow-up visits and cosmetic evaluations.
Measure: Number; unit: Incisions with good outcome
Arm/Group | Prineo | Suture
Number analyzed (Participants) | 60 | 60
Incisions with good outcome | 37 | 32
Statistical Analysis 1: Comparison: Prineo vs Suture; Test type: Superiority or Other; p = 0.2266, McNemar

5. Secondary Outcome: Cosmetic Outcome
Description: as for outcome 3
Time Frame: 12 months
Population: There were 59 participants who completed all follow-up visits and cosmetic evaluations.
Measure: Number; unit: Incisions with good outcome
Arm/Group | Prineo | Suture
Number analyzed (Participants) | 59 | 59
Incisions with good outcome | 40 | 43
Statistical Analysis 1: Comparison: Prineo vs Suture; Test type: Superiority or Other; p = 0.5078, McNemar

ADVERSE EVENTS:
Time Frame: 90+/-10 days following treatment
Description: Recorded as reported whether spontaneously volunteered or in response to questioning about well-being at all follow-up visits.
Groups:
- Procedure: On same patient, one breast is randomized to control and one breast is randomized to experimental arm. Patient is own control.
Arm/Group | Prineo | Suture | Procedure
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/79 | 2/79
Other Adverse Events (participants affected / at risk) | 31/79 | 21/79 | 50/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prineo (N=79) | Suture (N=79) | Procedure (N=79)
Elective Brachioplasty (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Subject underwent planned bilateral brachioplasty for hanging skin. The event required hospitalisation for medical/surgical intervention. In the opinion of the Investigator, the event was classified as not related to sutures or Prineo.
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Following treatment, patient experienced postoperative sepsis and was hospitalized. Patient required surgical reintervention and was treated with antibiotics. No action was taken with respect to the study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Prineo (N=79) | Suture (N=79) | Procedure (N=79)
Blistering (Skin and subcutaneous tissue disorders) | 8 (8) | 0/0 (0) | 5 (5)
Pain (General disorders) | 17 (17) | 15 (15) | 18 (18)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 2/78 (2) | 5 (5) — Itchiness at application site assessed as not related to device but to procedure.
Nausea (Gastrointestinal disorders) | 3 (3) | 2/78 (2) | 12 (12) — Nausea was assessed as not related to device but to procedure.
Hematoma (Vascular disorders) | 3 (3) | 1 (1) | 9 (9) — Events assessed as not related to device but to procedure.
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 4 (4) — Events assessed not related device but to procedure.
Procedure Pain (Injury, poisoning and procedural complications) | 6 (6) | 6 (6) | 16 (16)
Open Wound (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 6 (6)

LIMITATIONS AND CAVEATS:
Limitations of this study include the fact that the patient served as her own control. Additionally, as in many device studies, because of the obvious difference in the investigated and the control devices, blinding was limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less